CLINICAL TRIAL: NCT02638168
Title: Effects of Evening Dose of Immediate Release Methylphenidate on Sleep in Children With Attention Deficit Hyperactivity Disorder: A Randomized Placebo-controlled Pilot Study
Brief Title: Effects of Evening Dose of Immediate Release Methylphenidate on Sleep in Children With ADHD
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: challenge in recruitment
Sponsor: Milton S. Hershey Medical Center (Other)
Collaborators: Children's Miracle Network (Other)
Responsible Party: Principal Investigator, Raman Baweja, Assistant Professor, Milton S. Hershey Medical Center
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: STUDY00003056
Record Dates: First submitted 2015-12-15; First posted 2015-12-23 (Estimated); Results first posted 2019-09-17 (Actual); Last update posted 2019-09-17 (Actual); Status verified 2019-09

CONDITIONS: Attention Deficit Disorder With Hyperactivity; Behavioral Insomnia of Childhood
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Immediate Release Methylphenidate (Active Comparator): With-in subjects trial. Subjects will be randomized to 0.3 mg/kg of Immediate Release Methylphenidate versus placebo over 3-weeks duration
  Interventions: Drug: Immediate Release Methylphenidate
- Placebo (Placebo Comparator): inert placebo ingredient
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Immediate Release Methylphenidate — The medication assessment procedure will be a double-blind, within-subject evaluation of placebo and matching evening dose of IR MPH rounded to the nearest 2.5mg increment with a max IR MPH dose of 0.3mg/kg. Expected evening dose range will be from 2.5mg to 20mg with most participants receiving between 5 to 15mg per evening dose. Dose will be determined based on current dose of their morning extended release stimulant
  Other Names: Generic Methylphenidate
  Arms: Immediate Release Methylphenidate
Drug: Placebo — inert placebo ingredient
  Arms: Placebo

SUMMARY:
Over 10% of children in the United States are diagnosed with ADHD, and nearly half of these children have moderate to severe impairments in sleep, further exacerbating their already impaired academic, emotional and social functioning. In children with ADHD, 34% of prescribed sleep medications are antipsychotics that can cause marked weight gain and metabolic changes; alternate medications have either been found to be ineffective, difficult to tolerate or are largely unstudied in youth. Delayed sleep onset is strongly correlated with active symptoms of ADHD and Oppositional Defiant Disorder (ODD), suggesting that better control of disruptive behaviors could improve sleep patterns and this application will assess if the extension of the therapeutic effects of CNS stimulants into the early evening improves sleep onset.

DETAILED DESCRIPTION:
The goal of this application is to assess the impact of safer treatment option Methylphenidate (MPH) on sleep and behavior problems in children with Attention Deficit Hyperactivity Disorder (ADHD) and Behavioral Insomnia of Childhood (BIC). ADHD affects over 11% of school-aged youth. Similarly, pediatric sleep disorders occur in over a third of children and impact multiple domains of the child's functioning as well as that of their parents. Children with ADHD are at an increased risk for sleep problems with a staggering comorbidity of up to 70%, while sleep deprivation worsens the already impaired social, emotional and academic functioning of children with ADHD. Therefore, improving sleep may translate into enhanced functioning in multiple realms. Delayed sleep onset latency (SOL) and bedtime resistance, the key component of the limit setting type of BIC, are particularly likely to occur in children with ADHD. Medications are commonly used for both conditions with over 6% of all school-aged children in the United States prescribed medication for ADHD and 7% for sleep. In children with ADHD, 34% of prescribed sleep medications are antipsychotics that can cause marked weight gain and metabolic changes. Alternate medications for sleep have either been found to be ineffective, difficult to tolerate or are largely unstudied in youth. MPH has an extensive database supporting their safety and efficacy. Objective sleep studies of MPH have not found consistent results, with a few studies reporting delayed SOL and while others report improved quality of sleep. Therefore, this proposal will evaluate the impact of extending MPH treatment into the early evening on sleep onset using a 3-week with-in subjects randomized trial of .3mg/kg of immediate release (IR) MPH dosed 3 hours before bedtime vs. placebo in 38 children with ADHD and chronically delayed SOL who have a history of prolonged stimulant usage. The investigators will recruit 38 children ages 6-12 of any gender and racial/ethnic status with ADHD who have been treated with stable morning dose of extended release (ER) MPH for an extended time period (30 days or more) from the primary care and psychiatry clinics at Hershey Medical Center in Hershey, PA. Recruitment will be split into three waves (13, 13, 12 participants). Parents will be reminded to administer the blinded medication dose by text message each evening (or phone call by study staff) 3 hours prior to the desired bedtime. Sleep onset will be measured by actigraphy and sleep log, with parents also reporting on level of ODD and ADHD symptoms in the evening.

ELIGIBILITY:
Inclusion Criteria:

1. Ages 6-12 (inclusive), and able to swallow capsule
2. Children who have been treated with a stable morning dose of Extended Release Methylphenidate or twice daily dose of Immediate Release Methylphenidate for an extended period of time (30 days or longer).
3. DSM V diagnosis of Attention Deficit Hyperactivity Disorder (ADHD): Diagnosis will be assessed on the NIMH Computerized Diagnostic Interview Schedule for Children (C-DISC), and parent and teacher rating scales.
4. Children with any ADHD subtype meeting the above criteria will be eligible, although, it is expected that the majority will be of the combined subtype of ADHD given the associate between this subtype and ODD symptoms. A diagnosis of any of the two Behavioral Insomnia of Childhood (BIC) subtypes associated with delayed SOL (limit setting or combined type) will be required.
5. Sex: male or female
6. Fluent in written and spoken English.

Exclusion Criteria:

1. Age < 6 years of age or >12 years of age.
2. Children who have not had Methylphenidate (Extended Release) treatment for an extended period of time (30 days or longer).
3. A diagnosis or suspicion of sleep-disordered breathing will be exclusionary as it is not expected to be impacted by Immediate Release Methylphenidate treatment.
4. Current psychotropics other than Methylphenidate (Extended Release or Immediate Release Methylphenidate). Children prescribed alpha agonists for adjunctive control of ADHD in combination with a MPH product will be allowed to enroll as long as they meet all other entry criteria (i.e. sleep must remained impaired with use of alpha agonist).
5. Regular use of other medications that impact sleep within the last 14 days (i.e.: sedating antihistamines, melatonin).
6. Active medical/psychiatric conditions that impact sleep (i.e.: severe asthma, Autism Spectrum Disorder diagnosis, marked developmental delay, or mood/anxiety disorder).

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 3 (Actual)
Dates: Start 2016-01; Primary Completion 2018-06 (Actual); Study Completion 2018-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Raman Baweja, M.D., M.S., Principal Investigator — Milton S. Hershey Medical Center
Locations (1):
- Milton S Hershey Medical Center, Hershey, Pennsylvania, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo: inert placebo ingredient
  Placebo: inert placebo ingredient
  We have total 6 screening and recruited 3 patients for this study
Period: Overall Study
Arm/Group | Immediate Release Methylphenidate | Placebo
Started (This was with-in subject trial) | 3 | 0
Completed | 3 | 0
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- With-in Subjects Trial: Subjects were randomized to 0.3 mg/kg Immediate Release Methylphenidate va placebo over 3-weeks duration
Arm/Group | With-in Subjects Trial
Number analyzed (Participants) | 3
Age, Continuous [Mean (Full Range); unit: years] | 8.3 [8 to 10]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 3
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Sleep Onset Latency (SOL) as Reported on the Parent Completed Sleep Log
Description: Sleep onset latency is defines as duration of time in bed until sleep, as reported on the parent completed sleep log
Time Frame: 3 weeks
Measure: Mean (Full Range); unit: minutes
Arm/Group | With-in Subjects Trial
Number analyzed (Participants) | 3
minutes | 61.04 [23.1 to 114.51]

2. Secondary Outcome: Sleep Onset Latency (SOL), Defined as Time in Bed Until Sleep by Actigraphy
Description: Sleep onset latency is defines as duration of time in bed until sleep actigraphy
Time Frame: 3 weeks
Measure: Mean (Full Range); unit: minutes
Arm/Group | With-in Subjects Trial
Number analyzed (Participants) | 3
minutes | 37.81 [0 to 95]

3. Secondary Outcome: Pittsburgh Side Effects Rating Scale
Description: Pittsburgh Side Effects Rating Scale to evaluate adverse reactions to Methylphenidate Higher scores mean a worse outcome (more side effects with medication) This scales has 13 items, which are reported as None (0), Mild (1), Moderate (2) and Severe (3) Total score is calculated by summiting all items. Total Score Ranges (0-39)
Time Frame: 3 weeks
Measure: Mean (Full Range); unit: score on a scale
Arm/Group | With-in Subjects Trial
Number analyzed (Participants) | 3
score on a scale | 3.66 [3 to 5]

4. Secondary Outcome: Sleep Offset
Time Frame: 3 weeks
Measure: Mean (Full Range); unit: minutes
Arm/Group | With-in Subjects Trial
Number analyzed (Participants) | 3
minutes | 604 [580 to 675]

5. Secondary Outcome: Total Sleep Time
Time Frame: 3 weeks
Measure: Mean (Full Range); unit: minutes
Arm/Group | With-in Subjects Trial
Number analyzed (Participants) | 3
minutes | 492.45 [432 to 585]

6. Secondary Outcome: Wake After Sleep Onset (WASO)
Time Frame: 3 weeks
Measure: Median (Full Range); unit: minutes
Arm/Group | With-in Subjects Trial
Number analyzed (Participants) | 3
minutes | 73.81 [29 to 147]

7. Secondary Outcome: Sleep Efficiency
Time Frame: 3 weeks
Measure: Mean (Full Range); unit: percentage of time spent asleep in bed
Arm/Group | With-in Subjects Trial
Number analyzed (Participants) | 3
percentage of time spent asleep in bed | 81.45 [72.61 to 89.14]

8. Secondary Outcome: Number of Wakings
Time Frame: 3 weeks
Measure: Mean (Full Range); unit: Wakings
Arm/Group | With-in Subjects Trial
Number analyzed (Participants) | 3
Wakings | 22.81 [15 to 33]

9. Secondary Outcome: Length of Wakings
Time Frame: 3 weeks
Measure: Mean (Full Range); unit: minutes
Arm/Group | With-in Subjects Trial
Number analyzed (Participants) | 3
minutes | 3.28 [1.52 to 5.88]

10. Secondary Outcome: Night to Night Variability (Weekends & Weekdays) - in Sleep Onset Latency Measured by Actigraphy
Description: We calculated Night to night variability by the difference between the mean sleep onset latency during the weekend days and the mean sleep onset latency during the weekdays.
Time Frame: 3 weeks
Measure: Mean (Full Range); unit: minutes
Arm/Group | With-in Subjects Trial
Number analyzed (Participants) | 3
minutes | 35.96 [0 to 95]

11. Secondary Outcome: Parent Rated 10-item IOWA
Description: Higher scores mean severe symptoms This scales has 10 items, which are reported as Not at all (0), just a little (1), pretty much (2) and very much (3) Total score is calculated by summiting all items. Total Score Ranges (0-30)
Time Frame: 3 weeks
Measure: Mean (Full Range); unit: score on a scale
Arm/Group | With-in Subjects Trial
Number analyzed (Participants) | 3
score on a scale | 13.3 [9 to 17]

12. Secondary Outcome: Affective Reactivity Index (ARI)
Description: Higher scores mean a worse symptoms This scales has 7 items, which are reported as Not true (0), somewhat true (1) certainly true (2) Total score is calculated by summiting all items. Total Score Ranges (0-14)
Time Frame: 3 weeks
Measure: Mean (Full Range); unit: score on a scale
Arm/Group | With-in Subjects Trial
Number analyzed (Participants) | 3
score on a scale | 5 [1 to 10]

ADVERSE EVENTS:
Time Frame: Over the 3 weeks during randomization trial
Arm/Group | With-in Subjects Trial
All-Cause Mortality (participants affected / at risk) | 0/3
Serious Adverse Events (participants affected / at risk) | 0/3
Other Adverse Events (participants affected / at risk) | 0/3

LIMITATIONS AND CAVEATS:
Only 3 participants were randomized.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-10-19): https://cdn.clinicaltrials.gov/large-docs/68/NCT02638168/Prot_SAP_000.pdf